CLINICAL TRIAL: NCT03888157
Title: A Multi-centre, Prospective, Non-interventional Study Investigating the Effect of Victoza® in Patients With Type 2 Diabetes in Iran Followed in a Real World Setting
Brief Title: A Research Study Looking at How Victoza® Works in People With Type 2 Diabetes in Iran, Followed in Local Clinical Routine
Acronym: VIEW-Iran
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4438; U1111-1213-4238 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-03-11; First posted 2019-03-25 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liraglutide: Patients with type 2 diabetes in Iran are to receive Victoza® for 26 weeks.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Patients will be treated according to the Iranian label for Victoza®, following routine clinical practice and at the discretion of the study doctor. The study doctor will determine the intended maintenance dose of Victoza®, as well as any changes to the maintenance dose thereafter. Patients will be treated according to the Iranian label for Victoza®, following routine clinical practice and at the discretion of the study doctor. The study doctor will determine the intended maintenance dose of Victoza®, as well as any changes to the maintenance dose thereafter. The physician's decision to initiate treatment with Victoza® is clearly separate from the opportunity to include the patient in the study.
  Other Names: Victoza®

SUMMARY:
The purpose of the study is to collect information on how the medicine Victoza® (liraglutide) works in people with Type 2 diabetes in Iran. Patients will get Victoza® as prescribed to them by their study doctor. The study will last for about 5 to 8 months. Patients will be asked to complete some questionnaires about their health and diabetes treatment. Patients will complete these during their normally scheduled visits with study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* The decision to initiate treatment with commercially available Victoza® has been made by the patient and the treating physician before and independently from the decision to include the patient in this study
* Patients diagnosed with type 2 diabetes mellitus (T2DM), with treatment planned according to the Iranian label for Victoza® at treatment initiation
* Available glycated haemoglobin A1c (HbA1c) value less than or equal to 12 weeks prior to initiation of treatment with Victoza®

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Known or suspected hypersensitivity to Victoza® or related products
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with T2DM in Iran judged by the study doctor for whom Victoza® is indicated are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin A1c (HbA1c) (percentage) | Week 0, week 26
  Measured in percentage.
Change in HbA1c (mmol/mol) | Week 0, week 26
  Measured in mmol/mol.

SECONDARY OUTCOMES:
Change in body weight (kilogram) | Week 0, week 26
  Measured in kilogram.
Change in body weight (percentage) | Week 0, week 26
  Measured in percentage.
Change in waist circumference | Week 0, week 26
  Measured in centimetres.
Change in fasting blood glucose (FBG) (self-measured) | Week 0, week 26
  Measured in mg/dL.
Change in total cholesterol (TC) | Week 0, week 26
  Measured in mg/dL.
Change in low density lipoprotein cholesterol (LDL-C) | Week 0, week 26
  Measured in mg/dL.
Change in high density lipoprotein cholesterol (HDL-C) | Week 0, week 26
  Measured in mg/dL.
Change in triglyceride (TG) | Week 0, week 26
  Measured in mg/dL.
Change in free fatty acid (FFA) | Week 0, week 26
  Measured in mg/dL.
Number of patients permanently discontinuing treatment with Victoza® | Week 26
  Number of patients.
Reasons for permanent treatment discontinuations | Week 26
  Number of occurrence of pre-specified events.
Changes in quality of life (EQ-5D index score) | Week 0, week 26
  Quality of life will be measured with the EQ-5D-5L instrument's index score. The EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems and extreme problems). The outcome will be presented as EQ-5D index values using the United Kingdom (UK) value set.
Changes in quality of life (EQ VAS) | Week 0, week 26
  Quality of life will be measured by EQ-5D-5L instrument's EQ visual analogue scale (EQ VAS). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. The scale is numbered from 0 to 100, where 0 indicates "worst" and 100 indicates "best". The outcome will be presented as EQ-5D VAS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (16):
- Iran (16):
  - Novo Nordisk Investigational Site, Ahvāz
  - Novo Nordisk Investigational Site, Ardabil
  - Novo Nordisk Investigational Site, Babol
  - Novo Nordisk Investigational Site, Gorgan
  - Novo Nordisk Investigational Site, Hamadan
  - Novo Nordisk Investigational Site, Hormozgan
  - Novo Nordisk Investigational Site, Isfahan
  - Novo Nordisk Investigational Site, Islamshahr
  - Novo Nordisk Investigational Site, Karaj
  - Novo Nordisk Investigational Site, Kerman
  - Novo Nordisk Investigational Site, Mashahd
  - Novo Nordisk Investigational Site, Mashhad
  - Novo Nordisk Investigational Site, Sari
  - Novo Nordisk Investigational Site, Shiraz
  - Novo Nordisk Investigational Site, Tehran
  - Novo Nordisk Investigational Site, Yazd

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results